CLINICAL TRIAL: NCT03963973
Title: A Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetic (PK) Profile of Multiple Oral Doses of RDN-929 in Healthy Older Adults
Brief Title: A 28 Day Parallel Group Study to Assess the Effects of RDN-929
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Participants no longer receiving intervention
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RDN-929-103
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDN-929 (Experimental): low, medium and high dose of RDN-929 capsules
  Interventions: Drug: RDN-929 oral capsule
- Placebo (Placebo Comparator): Matching placebo capsules
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: RDN-929 oral capsule — low, medium and high dose
  Arms: RDN-929
Drug: Placebo oral capsule — matching placebo dose
  Arms: Placebo

SUMMARY:
Eligibility will be assessed during a screening period of up to 4 weeks. Subjects will take study medication once daily up to and including Day 28. Safety, tolerability and PK will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or postmenopausal or surgically sterile females age 55 - 85 years old.
* Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and ECG recording

Exclusion Criteria:

* Any history of major psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal (ULN)
* A clinically significant abnormality on physical examination, neurological examination, ECG, or laboratory evaluations
* A clinically significant vital signs abnormality, as judged by the principal investigator

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 9 weeks
  Screening to end of study, up to 9 weeks
Number of subjects with Physical exam findings | up to 9 weeks
  Screening to end of study, up to 9 weeks
Number of subjects with Clinical safety lab changes | up to 9 weeks
  Screening to end of study, up to 9 weeks
Number of subjects with Systolic blood pressure changes | up to 9 weeks
  Screening to end of study, up to 9 weeks
Number of subjects with Heart rate changes | up to 9 weeks
  Screening to end of study, up to 9 weeks
Number of subjects with 12 Lead ECG changes | up to 9 weeks
  Screening to end of study, up to 9 weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration, Cmax | Day 1 to Day 28
  RDN-929 and primary metabolite ROD-1610
Area Under the plasma and CSF concentration time curve, AUC | Day 1 to Day 28
  RDN-929 and primary metabolite ROD-1610

CONTACTS AND LOCATIONS:
Overall Officials: PI, Principal Investigator — QPS Holdings LLC
Locations (2):
- Netherlands (2):
  - Brain Research Center, Amsterdam
  - QPS Netherlands B.V., Leeuwarden

IPD SHARING:
Plan to Share IPD: No